CLINICAL TRIAL: NCT01499628
Title: Eccentric Fixation From Enhanced Clinical Training (EFFECT): A Randomised Clinical Trial for Patients With AMD
Brief Title: EFFECT:Eccentric Fixation From Enhanced Clinical Training
Acronym: EFFECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Moorfields Eye Hospital NHS Foundation Trust (Other)
Collaborators: British Eye Research Foundation, operating as Fight for Sight (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RUBG1008; Fight for Sight Ref: 1777/78 (Other Grant/Funding Number: Funder)
Record Dates: First submitted 2011-12-20; First posted 2011-12-26 (Estimated); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Age Related Macular Degeneration (ARMD)
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1-Control (No Intervention): No extra training will be given.
- Group 2-Control plus supervised reading (Active Comparator): The same amount of contact time as Groups 3 and 4 - three 45 minute sessions completed over three weeks.
  Interventions: Behavioral: Supervised Reading
- Group 3-EVT at the PRL (Experimental): Eccentric viewing training at the Preferred Retinal Locus (PRL), using reading/target cards. Three 45 minute sessions completed over three weeks.
  Interventions: Behavioral: EVT at the PRL
- Group 4-EVT at the TRL (Experimental): Eccentric viewing training at the Trained Retinal Locus (TRL), using reading/target cards and microperimeter. Three 45 minute sessions completed over three weeks.
  Interventions: Behavioral: EVT at the TRL

INTERVENTIONS:
Behavioral: Supervised Reading — Participant attends once a week for three weeks for a 45 minute appointment of supervised reading using appropriate spectacles and/or glasses
  Arms: Group 2-Control plus supervised reading
Behavioral: EVT at the PRL — Eccentric viewing training at the Preferred Retinal Locus (PRL), using reading/target cards. Three 45 minute sessions completed over three weeks.
  Arms: Group 3-EVT at the PRL
Behavioral: EVT at the TRL — Participant attends once a week for three weeks for a 45 minute appointment of TRL training using the MAIA microperimeter and then further reading using magnifiers and/or spectacles.
  Arms: Group 4-EVT at the TRL

SUMMARY:
Age-related macular degeneration (AMD) is the leading cause of severe visual impairment in the UK, Europe and N America. Low vision patients with AMD have great difficulty reading, which leads to a loss of independence and reduced quality of life. Magnifiers alone do not compensate for loss of central vision in AMD. It has been proposed that special low vision training can improve reading ability in patients with AMD. Training programmes are widely available in the US and Scandinavia, but not in the UK, partly because there is a lack of evidence from Randomised Control Trials (RCT) showing that they are effective. The investigators are conducting a clinical trial comparing the conventional hospital-based low vision service to enhanced rehabilitation programmes that include Eccentric Viewing training. Eccentric viewing training involves teaching patients who have lost their central vision to use a new area of retina for visual tasks. Patients are either taught to improve the use of the part of the retina they naturally start using after their central vision is lost, their so-called preferred retinal locus (PRL), or, alternatively, they are taught to use a different retinal area that is thought to be better suited for everyday visual tasks, the so-called trained retinal locus (TRL). The investigators plan to compare the two types of eccentric viewing training to conventional hospital-based low vision care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of age-related macular degeneration
* Visual acuity 6/12 to 3/60 inclusive in the better eye
* Dense central scotoma confirmed by microperimetry

Exclusion Criteria:

* Patients who are not fluent in English or are cognitively impaired
* Patients with serious hearing impairment
* Patients who are hospital inpatients, who are living in nursing homes or are otherwise non-independent
* Ocular co-morbidity (other than mild cataract) in the better eye
* Recent low vision assessment or eccentric viewing training

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-04-27 (Actual); Primary Completion 2015-11-26 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Score on the Massof Activity Inventory - 6 month follow up | Change from Baseline in Massof Activity Inventory at 6 month follow up

SECONDARY OUTCOMES:
Reading Speed (ReST) - Final Assessment | Change from Baseline in Reading Speed (ReST) at Final Assessment
Quality of Life (MacDQoL) - Final Assessment | Change from Baseline in Quality of Life (MacDQoL) at Final Assessment
Quality of Life (MacDQoL) - 6 month follow up | Change from Baseline in Quality of Life (MacDQoL) at 6 month follow up
Quality of Life (MacDQoL) - 12 month follow up | Change from Baseline in Quality of Life (MacDQol) at 12 month follow up
Self-reported health status (EQ-5D) - Final Assessment | Change from Baseline in EQ-5D score at Final Assessment
Self-reported health status (EQ-5D) - 6 month follow up | Change from Baseline in EQ-5D score at 6 month follow up
Self-reported health status (EQ-5D) - 12 month follow up | Change from Baseline in EQ-5D score at 12 month follow up
Time Trade Off (TTO) - 6 month follow up | Change from Baseline in Time Trade Off (TTO) score at 6 month follow up
WHO (Five) Well-Being Index (WBI-5) - Final Assessment | Change from Baseline in WBI-5 score at Final Assessment
WHO (Five) Well-Being Index (WBI-5) - 6 month follow up | Change from Baseline in WBI-5 score at 6 month follow up
WHO (Five) Well-Being Index (WBI-5) - 12 month follow up | Change from Baseline in WBI-5 score at 12 month follow up
Interpersonal Support Evaluation List (ISEL) - Final Assessment | Change from Baseline in Interpersonal Support Evaluation List (ISEL) at Final Assessment
Interpersonal Support Evaluation List (ISEL) - 6 month follow up | Change from Baseline in Interpersonal Support Evaluation List (ISEL) at 6 month follow up
Interpersonal Support Evaluation List (ISEL) - 12 month follow up | Change from Baseline in Interpersonal Support Evaluation List (ISEL) at 12 month follow up
Acceptance and Self Worth Adjustment Scale (AS-WAS) - Final Assessment | Change from Baseline in Acceptance and Self Worth Adjustment Scale (AS-WAS) at Final Assessment
Acceptance and Self Worth Adjustment Scale (AS-WAS) - 6 month follow up | Change from Baseline in Acceptance and Self Worth Adjustment Scale (AS-WAS) at 6 month follow up
Acceptance and Self Worth Adjustment Scale (AS-WAS) - 12 month follow up | Change from Baseline in Acceptance and Self Worth Adjustment Scale (AS-WAS) at 12 month follow up
Massof Activity Inventory - Final Assessment | Change from Baseline in Massof Activity Inventory at Final Assessment
Massof Activity Inventory - 12 month follow up | Change from Baseline in Massof Activity Inventory at 12 month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Gary S Rubin, PhD, Principal Investigator — University College, London
Locations (1):
- Moorfields Eye Hospital, London, United Kingdom